CLINICAL TRIAL: NCT01150890
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Efficacy of AMG 827 in Subjects With Moderate to Severe Crohn's Disease
Brief Title: Brodalumab (AMG 827) in Adults With Moderate to Severe Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early based on an imbalance in worsening Crohn's disease in active treatment groups
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20090072; 2010-019544-39 (EudraCT Number)
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Results first posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-11

CONDITIONS: Crohn's Disease
Keywords: Ileal Crohn's Disease; Ileo-colonic Crohn's Disease; Colonic Chron's Disease
MeSH Terms: conditions — Crohn Disease | interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo intravenously at baseline and week 4.
  Interventions: Drug: Placebo
- Brodalumab 210 mg (Experimental): Participants received 210 mg brodalumab intravenously at baseline and week 4.
  Interventions: Biological: Brodalumab
- Brodalumab 350 mg (Experimental): Participants received 350 mg brodalumab intravenously at baseline and week 4.
  Interventions: Biological: Brodalumab
- Brodalumab 700 mg (Experimental): Participants received 700 mg brodalumab intravenously at baseline and week 4.
  Interventions: Biological: Brodalumab

INTERVENTIONS:
Biological: Brodalumab — Administered as as an intravenous (IV) infusion over at least 30 minutes.
  Other Names: AMG 827
  Arms: Brodalumab 210 mg; Brodalumab 350 mg; Brodalumab 700 mg
Drug: Placebo — Administered as as an intravenous (IV) infusion over at least 30 minutes.
  Arms: Placebo

SUMMARY:
The study will examine the safety and effectiveness of brodalumab for the treatment of moderate to severe Crohn's disease. Participants will randomly assigned to receive either brodalumab or placebo (a lookalike liquid that doesn't have any drug in it) and neither the doctor nor the patient will know what treatment is being given.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ileal, ileo-colonic, or colonic Crohn's disease for a minimum of 6 months prior to initiating study drug
* Moderately to severely active Crohn's disease, as defined by a CDAI score >250 and < 450 at baseline
* Evidence of active inflammation

Exclusion Criteria:

* Short bowel syndrome
* Stricture with obstructive symptoms within 3 months
* Bowel surgery within 3 months
* Ileostomy and/or colostomy
* Any gastric or intestinal pouch
* Ulcerative colitis
* Evidence of an infected abscess
* Bowel perforation or evidence of noninflammatory obstruction during the 6 months
* Stool positive for C. Difficile toxin at screening
* Presence of active infection requiring treatment
* Serious infection within 8 weeks
* Significant concurrent medical conditions
* Pregnant or breast feeding
* Significant Laboratory abnormalities
* Any anti-tumor necrosis factor (TNF) agent within 2 months
* Steroid enemas within 2 weeks
* Tysabri (natalizumab) within 1 year
* Biologic agents (eg, ustekinumab), experimental procedures, or live vaccines within 3 months
* Cyclosporine, mycophenolate mofetil, sirolimus (rapamycin),thalidomide or tacrolimus within 2 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-11-09 (Actual); Primary Completion 2011-10-15 (Actual); Study Completion 2011-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (50):
- United States (18):
  - Research Site, Birmingham, Alabama
  - Research Site, Dothan, Alabama
  - Research Site, Lowell, Arkansas
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Hammond, Louisiana
  - Research Site, Chevy Chase, Maryland
  - Research Site, Rochester, Minnesota
  - Research Site, Mexico, Missouri
  - Research Site, Egg Harbor, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Germantown, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, San Antonio, Texas
  - Research Site, Logan, Utah
  - Research Site, Ogden, Utah
- Australia (4):
  - Research Site, Kurralta Park, South Australia
  - Research Site, Box Hill
  - Research Site, Fitzroy
  - Research Site, Fremantle
- Belgium (4):
  - Research Site, Bonheiden
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Roeselare
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- France (5):
  - Research Site, Lille
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Maastricht
  - Research Site, Rotterdam
- Poland (4):
  - Research Site, Bydgoszcz
  - Research Site, Olsztyn
  - Research Site, Opole
  - Research Site, Sopot
- Spain (4):
  - Research Site, Pontevedra, Galicia
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Barcelona
  - Research Site, Madrid

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 39 centers in Australia, Belgium, Canada, Spain, France, Netherlands, Poland, and the United States (US).
  A total of 212 subjects were screened and 130 participants were randomized.
Pre-assignment Details: After completing all screening assessments and meeting all eligibility criteria, participants were randomized in a 1:1:1:1 ratio to one of four treatment groups.
Period: Overall Study
Arm/Group | Placebo | Brodalumab 210 mg | Brodalumab 350 mg | Brodalumab 700 mg
Started | 32 | 32 | 33 | 33
Received Study Drug | 32 | 31 | 32 | 33
Completed (Completing the study is defined as completing 12 weeks of study evaluations) | 28 | 19 | 21 | 16
Not Completed | 4 | 13 | 12 | 17
Not completed — Other | 0 | 1 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Administrative Decision | 4 | 4 | 5 | 6
Not completed — Ineligibility determined | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Disease progression | 0 | 7 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Brodalumab 210 mg | Brodalumab 350 mg | Brodalumab 700 mg | Total
Number analyzed (Participants) | 32 | 32 | 33 | 33 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (13.0) | 32.8 (10.2) | 36.8 (12.6) | 36.7 (10.0) | 35.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 21 | 21 | 78
  Male | 15 | 13 | 12 | 12 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 25 | 26 | 26 | 27 | 104
  Unknown or Not Reported | 7 | 6 | 6 | 5 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 24 | 23 | 26 | 27 | 100
  Other | 1 | 1 | 1 | 1 | 4
  Unknown | 7 | 6 | 6 | 5 | 24
Predominant Location of Crohn's Disease (CD) Involvement [Count of Participants; unit: Participants]
  Ileal | 6 | 5 | 4 | 3 | 18
  Ileo-colonic | 17 | 19 | 17 | 16 | 69
  Colonic | 8 | 7 | 11 | 13 | 39
  Missing | 0 | 1 | 0 | 0 | 1
  Unknown | 1 | 0 | 1 | 1 | 3
Duration of Crohn's Disease [Mean (Standard Deviation); unit: years] — Population: Participants with available data
  years
    number analyzed (Participants) | 32 | 31 | 33 | 32 | 128
    (all) | 11.38 (9.35) | 9.57 (7.64) | 14.21 (10.35) | 11.71 (7.36) | 11.75 (8.84)
Crohn's Disease Activity Index (CDAI) [Mean (Standard Deviation); unit: score on a scale] — The CDAI measures the severity of active disease using 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). The CDAI score is calculated by summing weighted scores for each item. CDAI scores range from 0 to 600, with higher scores indicating greater disease activity. Population: Participants with available data
  score on a scale
    number analyzed (Participants) | 32 | 29 | 33 | 33 | 127
    (all) | 327.7 (63.0) | 333.2 (61.9) | 334.5 (60.3) | 315.4 (54.0) | 327.5 (59.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Remission at Week 6
Description: Clinical remission is defined by a CDAI score of ≤ 150 points. The CDAI measures the severity of active disease using 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). The CDAI score is calculated by summing weighted scores for each item. CDAI scores range from 0 to 600, with higher scores indicating greater disease activity.
Time Frame: Week 6
Population: The full analysis set included all randomized participants; missing data were analyzed using the non-responder imputation method.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brodalumab 210 mg | Brodalumab 350 mg | Brodalumab 700 mg
Number analyzed (Participants) | 32 | 32 | 33 | 33
percentage of participants | 3.1 | 3.1 | 15.2 | 9.1
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg vs Brodalumab 350 mg vs Brodalumab 700 mg; The primary null hypothesis was tested sequentially using a linear trend test at the significance level of 0.05 (two-sided) using logistic regression modeling; Test type: Superiority; p = 0.1941, Overall Trend test
Statistical Analysis 2: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 1.0000, Chi-squared; Difference in Response Rate = 0.0000, 95% CI 2-sided [-0.09 to 0.09]
Statistical Analysis 3: Comparison: Placebo vs Brodalumab 350 mg; Test type: Superiority; p = 0.0966, Chi-squared; Difference in Response Rate = 0.1203, 95% CI 2-sided [-0.02 to 0.26]
Statistical Analysis 4: Comparison: Placebo vs Brodalumab 700 mg; Test type: Superiority; p = 0.3208, Chi-squared; Difference in Response Rate = 0.0597, 95% CI 2-sided [-0.06 to 0.17]

2. Secondary Outcome: Percentage of Participants Who Achieved a CDAI Response at Week 6
Description: CDAI response is defined as a reduction from baseline in CDAI score of ≥ 100 points.
  The CDAI measures the severity of active disease using 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). The CDAI score is calculated by summing weighted scores for each item. CDAI scores range from 0 to 600, with higher scores indicating greater disease activity.
Time Frame: Week 6
Population: Full analysis set; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brodalumab 210 mg | Brodalumab 350 mg | Brodalumab 700 mg
Number analyzed (Participants) | 32 | 31 | 33 | 33
percentage of participants | 12.5 | 16.1 | 27.3 | 15.2
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.6831, Chi-squared; Difference in Response Rate = 0.0363, 95% CI 2-sided [-0.14 to 0.21]
Statistical Analysis 2: Comparison: Placebo vs Brodalumab 350 mg; Test type: Superiority; p = 0.1396, Chi-squared; Difference in Response Rate = 0.1477, 95% CI 2-sided [-0.04 to 0.34]
Statistical Analysis 3: Comparison: Placebo vs Brodalumab 700 mg; Test type: Superiority; p = 0.7588, Chi-squared; Difference in Response Rate = 0.0265, 95% CI 2-sided [-0.14 to 0.19]

3. Secondary Outcome: Change From Baseline in CDAI at Week 6
Description: The CDAI measures the severity of active disease using 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). The CDAI score is calculated by summing weighted scores for each item. CDAI scores range from 0 to 600, with higher scores indicating greater disease activity.
  A negative change from baseline indicates improvement.
Time Frame: Baseline and week 6
Population: Full analysis set; missing CDAI scores were imputed using baseline values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Brodalumab 210 mg | Brodalumab 350 mg | Brodalumab 700 mg
Number analyzed (Participants) | 32 | 29 | 33 | 33
score on a scale | -28.2 (86.0) | -8.7 (95.3) | -35.4 (105.6) | -0.6 (105.9)
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.4161, ANCOVA; Analysis of covariance (ANCOVA) model adjusted for baseline CDAI score
Statistical Analysis 2: Comparison: Placebo vs Brodalumab 350 mg; Test type: Superiority; p = 0.8094, ANCOVA; ANCOVA model adjusted for baseline CDAI score
Statistical Analysis 3: Comparison: Placebo vs Brodalumab 700 mg; Test type: Superiority; p = 0.3040, ANCOVA; ANCOVA model adjusted for baseline CDAI score

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical trial participant, including worsening of a pre-existing medical condition. The event does not necessarily have a causal relationship with study treatment. A treatment-emergent AE is an event that occurred after the initiation of study drug or was already present prior to the initiation of study drug but worsened in either intensity or frequency after the initiation of study drug.
  A serious AE is an adverse event that met at least one of the following criteria:
  * fatal,
  * life threatening,
  * required in-patient hospitalization or prolongation of existing hospitalization,
  * resulted in persistent or significant disability/incapacity,
  * congenital anomaly/birth defect, and/or
  * other significant medical hazard.
  The investigator assessed whether each AE was possibly related to the study drug.
Time Frame: From first dose of study drug up to week 12.
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Brodalumab 210 mg | Brodalumab 350 mg | Brodalumab 700 mg
Number analyzed (Participants) | 32 | 31 | 32 | 33
Participants
  All treatment emergent adverse events (TEAEs) | 25 | 23 | 27 | 28
  Serious adverse events | 2 | 3 | 8 | 9
  Fatal adverse events | 0 | 0 | 0 | 0
  TEAEs leading to discontinuation of study drug | 1 | 3 | 3 | 3
  TEAEs leading to discontinuation from study | 0 | 4 | 3 | 3
  Treatment-related treatment-emergent adverse events (TRTEAE) | 10 | 13 | 21 | 14
  Treatment-related serious adverse events | 0 | 3 | 4 | 5
  Treatment-related fatal adverse events | 0 | 0 | 0 | 0
  TRTEAE leading to discontinuation of study drug | 1 | 2 | 2 | 0
  TRTEAE leading to discontinuation from study | 0 | 2 | 2 | 0

5. Secondary Outcome: Maximum Observed Concentration (Cmax) of Brodalumab
Description: An optional pharmacokinetic (PK) substudy was offered to participants at a subset of sites and required additional informed consent.
  Serum concentrations of brodalumab were measured using a validated analytical method, enzyme-linked immusosorbent assay (ELISA). The lower limit of quantification (LLOQ) for the assay was 0.0500 μg/mL.
Time Frame: After first dose on Day 1 (pre-dose and within 15 minutes after the end of infusion [EOI]), day 4-6, 15, and 29 (pre-dose) and after second dose on day 29 (pre-dose and within 15 minutes after EOI), days 32-34, 43, 57, 64-66, and 85.
Population: The PK analysis set includes participants in the PK substudy who received at least one dose of brodalumab and who provided valid drug concentration data at each sampling time point in Weeks 1 to 4, or in Week 5 to 12, and for whom at least one PK parameter or endpoint could be adequately estimated.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Brodalumab 210 mg | Brodalumab 350 mg | Brodalumab 700 mg
Number analyzed (Participants) | 5 | 8 | 10
μg/mL
  After first dose | 53.1 (6.40) | 96.4 (17.6) | 184 (64.9)
  After second dose: number analyzed (Participants) | 3 | 6 | 4
  After second dose | 54.5 (1.08) | 98.7 (20.6) | 171 (63.2)

6. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Brodalumab
Description: as for outcome 5
Time Frame: as for outcome 5
Population: The PK analysis set with available data
Measure: Median (Full Range); unit: days
Arm/Group | Brodalumab 210 mg | Brodalumab 350 mg | Brodalumab 700 mg
Number analyzed (Participants) | 5 | 8 | 10
days
  After first dose | 0.034 [0.028 to 0.22] | 0.034 [0.021 to 0.050] | 0.036 [0.024 to 0.047]
  After second dose: number analyzed (Participants) | 3 | 6 | 4
  After second dose | 0.031 [0.026 to 0.039] | 0.033 [0.024 to 0.042] | 0.029 [0.024 to 0.039]

7. Secondary Outcome: Area Under the Serum Concentration Versus Time Curve, From Time Zero to the Last Measurable Concentration (AUClast) for Brodalumab
Description: as for outcome 5
Time Frame: as for outcome 5
Population: The PK analysis set with available data.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Brodalumab 210 mg | Brodalumab 350 mg | Brodalumab 700 mg
Number analyzed (Participants) | 5 | 8 | 10
day*μg/mL
  After first dose | 243 (61.0) | 501 (190) | 1428 (715)
  After second dose: number analyzed (Participants) | 3 | 6 | 4
  After second dose | 164 (124) | 622 (330) | 1558 (691)

8. Secondary Outcome: Area Under the Serum Concentration Versus Time Curve From Time Zero to 28 Days (AUC0-28) for Brodalumab
Description: as for outcome 5
Time Frame: After first dose on Day 1 (pre-dose and within 15 minutes after the end of infusion [EOI]), day 4-6, 15, and 29 (pre-dose) and after second dose on day 29 (pre-dose and within 15 minutes after EOI), days 32-34, 43, and 57.
Population: The PK analysis set with available data.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Brodalumab 210 mg | Brodalumab 350 mg | Brodalumab 700 mg
Number analyzed (Participants) | 5 | 8 | 10
day*μg/mL
  After first dose | 243 (61.0) | 501 (190) | 1432 (714)
  After second dose: number analyzed (Participants) | 3 | 6 | 4
  After second dose | 164 (124) | 595 (268) | 1434 (597)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to week 12.
Arm/Group | Placebo | Brodalumab 210 mg | Brodalumab 350 mg | Brodalumab 700 mg
Serious Adverse Events (participants affected / at risk) | 2/32 | 3/31 | 8/32 | 9/33
Other Adverse Events (participants affected / at risk) | 20/32 | 21/31 | 23/32 | 20/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | Brodalumab 210 mg (N=31) | Brodalumab 350 mg (N=32) | Brodalumab 700 mg (N=33)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 2 | 5 | 7
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | Brodalumab 210 mg (N=31) | Brodalumab 350 mg (N=32) | Brodalumab 700 mg (N=33)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 3 | 0
Abdominal tenderness (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Anal fistula (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 3 | 1 | 2 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 6 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 4
Proctalgia (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Fatigue (General disorders) | 1 | 1 | 1 | 2
Pyrexia (General disorders) | 4 | 3 | 8 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 4 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 2 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 1 | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 3
Viral infection (Infections and infestations) | 0 | 0 | 0 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 3 | 0
Headache (Nervous system disorders) | 5 | 1 | 2 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 4 | 1
Proteinuria (Renal and urinary disorders) | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.